CLINICAL TRIAL: NCT02156375
Title: A Phase 1, Randomized, Open-label, Parallel-design Study to Compare Single-dose Pharmacokinetics of Intravenous Ustekinumab Delivered in 2 Different Liquid in Vial Formulations
Brief Title: A Pharmacokinetic Study of Single-Dose Intravenous Ustekinumab Delivered in 2 Different Liquid in Vial Formulations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR104186; CNTO1275NAP1002
Record Dates: First submitted 2014-06-03; First posted 2014-06-05 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-03

CONDITIONS: Healthy
Keywords: Healthy; Ustekinumab; STELARA®
MeSH Terms: interventions — Ustekinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ustekinumab 90 mg/mL (Experimental)
  Interventions: Drug: Ustekinumab
- Ustekinumab 5 mg/mL (Experimental)
  Interventions: Drug: Ustekinumab

INTERVENTIONS:
Drug: Ustekinumab — Participants will receive a single 6 milligram per kilogram (mg/kg) intravenous infusion of 90 milligram per milliliter (mg/mL) liquid in vial (LIV) formulation, diluted in saline, on Day 1.
  Other Names: STELARA®
  Arms: Ustekinumab 90 mg/mL
Drug: Ustekinumab — Participants will receive a single 6 mg/kg intravenous infusion of 5 mg/mL LIV formulation, diluted in saline, on Day 1.
  Other Names: STELARA®
  Arms: Ustekinumab 5 mg/mL

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetic (PK) (blood levels) comparability of 2 different formulations of ustekinumab, 90 milligram per milliliter (mg/mL) liquid in vial (LIV) and 5 mg/mL LIV, following a single intravenous administration of 6 milligram per kilogram (mg/kg) ustekinumab, diluted in saline, in healthy participants.

DETAILED DESCRIPTION:
This is a multicenter (when more than one hospital or medical school team work on a medical research study), randomized (study drug is assigned by chance), parallel (a clinical trial comparing the response in two or more groups of participants receiving different treatments), open-label (all people know the identity of the intervention) single-dose, inpatient/outpatient study in healthy participants. The study consists of following periods: Screening (within 28 days before study drug administration), inpatient period (Day 1 to 4) and outpatient period (up to Day 141). Eligible participants will be randomly assigned in a 1:1 ratio to either 1 of 2 treatment groups (that is, Ustekinumab 90 mg/mL or Ustekinumab 5 mg/mL) and will receive treatment on Day 1. The PK comparability of 2 different formulations of ustekinumab, diluted in saline, will be evaluated primarily. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Have a weight in the range of 50.0 kilogram (kg) to 90.0 kg, inclusive and a body mass index (BMI) of 18.5 kilogram per square meter (kg/m^2) to 29.0 kg/m^2, inclusive
* If a woman, she must be incapable of pregnancy or using a highly effective method of birth control
* A woman must have a negative serum pregnancy test
* A man who is sexually active with a woman of childbearing potential and has not had a vasectomy must agree to use a barrier method of birth control
* Participant must be willing and able to adhere to the prohibitions and restrictions specified in this protocol
* Are nonsmokers or agree to smoke no more than 10 cigarettes or 2 cigars per day throughout the study

Exclusion Criteria:

* Participant currently has or has a history of any clinically significant medical illness or medical disorders including malignancy
* Participant has previously received ustekinumab
* Participant has a known or suspected intolerance or hypersensitivity to any biologic medication including ustekinumab
* Participant has received an investigational drug within a specified period prior to the planned first dose of study drug or is currently enrolled in an investigational study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2014-05; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | Day 0 through Day 113
  The Cmax is the maximum observed plasma concentration of study drug.
Area under the serum concentration versus time curve from time zero to infinity (AUC[0-inf]) | Day 0 through Day 113
  The AUC(0-inf) is the area under the serum concentration versus time curve from time zero to infinity with extrapolation of the terminal phase.

SECONDARY OUTCOMES:
Number of participants with adverse events (AEs) and serious adverse events (SAEs) | Baseline up to Day 141
  An AE is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non investigational) product and does not necessarily have a causal relationship with the treatment. An SAE is any untoward medical occurrence that meets any of the following conditions: results in death, is life threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, or is a congenital anomaly/birth defect.
Area under the serum concentration versus time curve from time zero to the time corresponding to the last quantifiable concentration (AUC[0-last]) | Day 0 through Day 113
  The AUC(0-last) is the area under the serum concentration versus time curve from time zero to the time corresponding to the last quantifiable concentration.
Terminal half-life (T1/2) | Day 0 through Day 113
  The T1/2 is the terminal half-life, that is, time required for the plasma concentration to decrease by one half.
Total systemic clearance (CL) | Day 0 through Day 113
  The CL is a quantitative measure of the rate at which a drug substance is removed from the body.
Volume of distribution (Vz) | Day 0 through Day 113
  The Vz is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug.
Number of participants with antibodies to ustekinumab | Baseline, Days 57 and 113
  Number of participants with antibodies to ustekinumab (tested using a validated immunoassay method) will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (3):
- United States (3):
  - Tempe, Arizona
  - Lincoln, Nebraska
  - Neptune City, New Jersey